CLINICAL TRIAL: NCT00549692
Title: Minimization, Double-blind, Placebo-controlled, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of Omega-3 Fatty Acids(Omacor®) for the Treatment of IgA Nephropathy
Brief Title: Efficacy and Safety of Omega-3 Fatty Acids(Omacor®) for the Treatment of Immunoglobulin A Nephropathy
Acronym: IgAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Collaborators: Pronova BioPharma ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-OM-8301
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omacor (Experimental)
  Interventions: Drug: Omega-3 fatty acid ethylester90
- Placebo Omacor (Placebo Comparator)
  Interventions: Drug: Omega-3 fatty acid ethylester90

INTERVENTIONS:
Drug: Omega-3 fatty acid ethylester90 — Dosage form :1g soft capsule Dosage : two capsules, twice a day.
  Other Names: Omacor®

SUMMARY:
The purpose of this study is to compare omega-3 fatty acids with placebo for efficacy in retardation of increase of serum creatinine(SCr) in IgA Nephropathy

DETAILED DESCRIPTION:
In the current clinical study, attempts are made to assess the safety and efficacy of omega-3 fatty acids by comparing between omega-3 fatty acids and the placebo in Korean patients with IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes age 18 or above
* Biopsy-proven IgA nephropathy
* Baseline serum creatinine ≥ 1.2mg/dl(Female),≥ 1.4mg/dl(Male)
* Able to give written informed consent

Exclusion Criteria:

* Hypertension SBP>160mmHg and/or DBP>100mmHg
* Subject, who in the investigator's opinion, has a systemic disease that would contraindicate participation in this study
* Use of omega-3 fatty acids or analog supplement
* Pregnancy or breast feeding at time of entry or unwillingness to comply with measures for contraception
* Current or recent (within 30 days) exposure to any investigational drug
* Subject who has hypersensitivity to this agent as a previous illness
* Low platelet(<100,000/㎕) or the subject who has a high risk of bleeding
* Use of corticosteroid during the treatment period or less than 3 months prior to the screening
* Use of anticoagulant during the treatment period or within 1 month or 6 half lives prior to screening
* Subject who in the investigator's opinion, would be confronted with a difficulty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-11; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The rate of number of patients that 50% or more increase in SCr after 42 months | 42 months

SECONDARY OUTCOMES:
The rate of number of patients that 50% or more increase in SCr after 6, 12, 24 and 36 months | 42 months
Mean change of SCr, estimated GFR, urine Protein/Creatinine ratio, urine Albumin/Creatinine ratio, serum Cystatin C, Lipid profile | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Suhnggwon Kim, Professor, Study Chair — Seoul National University Hospital; Byung-Joo Park, MD,PhD,FISPE, Principal Investigator — Seoul National University College of Medicine
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kyhung Hee University medical center, Seoul
  - Samsumg Medical Center, Seoul
  - Kangnam St. May's Hospital, Seoul